CLINICAL TRIAL: NCT03380195
Title: Effects of Watermelon Juice on Heart Rate Recovery and Post-exercise Muscle Soreness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2487100
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Heart Rate Recovery
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Watermelon juice (Experimental)
  Interventions: Other: Watermelon juice
- Sport drink (Active Comparator)
  Interventions: Other: Sport drink
- Sugar water (Active Comparator)
  Interventions: Other: Sugar water
- Water (Placebo Comparator)
  Interventions: Other: Water

INTERVENTIONS:
Other: Watermelon juice — Subject drinks 355ml of watermelon juice 1 hour prior to submaximal exercise
  Arms: Watermelon juice
Other: Sport drink — Subject drinks 355ml of Gatorade 1 hour prior to submaximal exercise
  Arms: Sport drink
Other: Sugar water — Subject drinks 355ml of sugar water (22.5g) 1 hour prior to submaximal exercise
  Arms: Sugar water
Other: Water — Subject drinks 355ml of water 1 hour prior to submaximal exercise
  Arms: Water

SUMMARY:
The purpose of this study was to determine the effects of a pre-exercise, single practical dose of watermelon juice, Gatorade, sugar water or water on heart rate recovery, blood lactate levels, and 24-hour post exercise muscle soreness.

ELIGIBILITY:
Inclusion Criteria:

* ages of 21-50 healthy adults

Exclusion Criteria:

* Suffering from injury
* Chronic inflammatory conditions
* Required dietary supplement use
* Required medication which affects blood pressure
* Smoking
* Pregnant woman
* Allergy to watermelon

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of heart rate after submax exercise | Baseline and every minute post exercise for a maximum 20 minutes post exercise.
  The participants then were fitted to cycling shoes and familiarized with the Lode cycle ergometer (Lode Excalibur Sport, Groningen, Netherlands), completed a warm-up and were asked to perform a criterion work rate trial ending at 80% predicted HRmax. Heart rate was recorded every minute post exercise for a maximum of 20 minutes post exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided